CLINICAL TRIAL: NCT01384786
Title: The Incidence of Thyroid Cancer in 4474 Patients Treated for Hyperthyroidism or Goiter
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Birte Nygaard md PhD, dept of endocinology O 106
Other Study IDs: JCEM070948
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Hyperthyreosis and Goiter; Thyroid Cancer
MeSH Terms: conditions — Goiter; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients with hyperthyroidism and/or goiter are evaluated with blood samples and scintiscan before they are treated with radioiodine for their thyroid disease. Because the investigators do not get a histologically/final diagnosis the investigators want to make sure, that the patients treated do not have a thyroid cancer when treated.

The investigators have found that thyroid cancer is not overlooked.

ELIGIBILITY:
Inclusion Criteria:

* all patients treated with radioiodine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Radioiodine treated patients
Sampling Method: Probability Sample
Enrollment: 4474 (Actual)
Dates: Start 2004-10; Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Vej-Hansen, Study Chair — Herlev Hospital, Copenhagen, Denmark
Locations (1):
- herlev Hospital, Copenhagen, Denmark